CLINICAL TRIAL: NCT02314351
Title: Intravenous Metoclopramide in the Acute Treatment of Migraine: A Double-blind, Randomized, Placebo-controlled Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Nurettin Özgür Doğan, M.D., Associate Professor, Kocaeli University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KOU KAEK 2014/315
Record Dates: First submitted 2014-12-05; First posted 2014-12-11 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2017-01

CONDITIONS: Migraine Disorders
Keywords: migraine disorders; migraine with aura; migraine without aura; pain management; emergency department
MeSH Terms: conditions — Migraine Disorders; Migraine with Aura; Migraine without Aura; Agnosia; Emergencies | interventions — Metoclopramide; Saline Solution; Fentanyl

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intravenous metoclopramide (Active Comparator): Intravenous metoclopramide, 10 mg (2 mL) in 98 mL 0.9% normal saline solution (total 100 mL)
  Interventions: Drug: Metoclopramide 10 mg; Drug: Placebo; Drug: Fentanyl
- Placebo (Placebo Comparator): 0.9% normal saline solution (total 100 mL)
  Interventions: Drug: Metoclopramide 10 mg; Drug: Placebo; Drug: Fentanyl

INTERVENTIONS:
Drug: Metoclopramide 10 mg — Intravenous form of metoclopramide is in the same appearance with placebo
  Other Names: Metoclopramide 10 mg (2 mL) in 100 mL normal saline
Drug: Placebo — Intravenous form of metoclopramide is in the same appearance with placebo
  Other Names: 100 mL normal saline
Drug: Fentanyl — Intravenous fentanyl (1 mcg/kg), if pain persists at 30th minute
  Other Names: Intravenous fentanyl

SUMMARY:
Migraine attacks were frequently diagnosed in the emergency departments. Also intravenous metoclopramide was a commonly used drug in the acute abortive treatment of migraine. However, the role of metoclopramide was based on three randomized, placebo-controlled studies, which were carried out with relatively few patients. Those trials suggested that metoclopramide produced larger improvements in visual analog scale (VAS) scores, however they revealed conflicting results and had significant methodological problems (risk of bias, allocation of concealment, intention-to-treat analysis). The investigators aimed to analyse the effects of intravenous metoclopramide in acute migraine attacks comparing with placebo.

ELIGIBILITY:
Inclusion Criteria:

* Presenting to the emergency department with migraine attack (with aura or without aura, according to International Headache Society criteria, 2013)
* The patients older than 18 years
* Patients who agree to participate to the study by reading and signing the informed consent document

Exclusion Criteria:

* The patients younger than 18 years
* Pregnants
* Patients taking any analgesic drugs last 2 hours
* Documented or declared allergy to metoclopramide
* Patients who are hemodynamically unstable
* Patients who do not agree to participate to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2014-12; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
The difference between pain scores for both drugs | 15th and 30th minutes
  The difference between pain scores (10- point numeric rating scale score) for metoclopramide and placebo groups

SECONDARY OUTCOMES:
Nausea and vomiting | 30th minute
  Change in nausea/vomiting status of the participants
Adverse reactions | 30th minute
  Number of participants with adverse events
Need for rescue analgesic | 30th minute
  Number of patients needed rescue analgesic at 30th minute
Change in the headache intensity | Between 24th and 72th hours
  Change in the headache intensity
Duplicative presentation to the emergency department | Between 24th and 72th hours
  With telephone call

CONTACTS AND LOCATIONS:
Overall Officials: Nurettin Özgür Doğan, Assoc. Prof, Principal Investigator — Kocaeli University, Faculty of Medicine
Locations (1):
- Kocaeli University, Faculty of Medicine, Köseköy, Kocaeli, Turkey (Türkiye)